CLINICAL TRIAL: NCT03365154
Title: Feasibility Clinical Trial of the Cardio Flow FreedomFlow Orbital Atherectomy System to Treat Peripheral Artery Disease
Brief Title: Feasibility Clinical Trial of the Cardio Flow Orbital Atherectomy System to Treat Peripheral Artery Disease (PAD)
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardio Flow, Inc. (Industry)
Collaborators: Libra Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010-031
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Artery Disease; Atherectomy; Orbital Atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Group (Experimental): Patients with occlusive arterial disease who meet the study criteria and provide informed consent will receive atherectomy treatment with the investigational device.
  Interventions: Device: Cardio Flow FreedomFlow™ Orbital Atherectomy System treatment; Device: Balloon Angioplasty

INTERVENTIONS:
Device: Cardio Flow FreedomFlow™ Orbital Atherectomy System treatment — Occlusive lesions will be treated using atherectomy with or without adjunctive low pressure balloon angioplasty.
  Other Names: Orbital Atherectomy Treatment
Device: Balloon Angioplasty — Low pressure balloon angioplasty may be used following atherectomy

SUMMARY:
This trial is a First in Human early feasibility study of a novel atherectomy device to treat peripheral artery disease. The trial is a prospective, single arm design that will enroll 10 patients at 1 - 2 sites. Patients will be followed at 30 days and 6 months to evaluate vessel patency following treatment. Safety will be assessed by monitoring adverse events throughout the study. Safety and Efficacy will be evaluated by comparing study results to established performance criteria,

DETAILED DESCRIPTION:
Feasibility Clinical Trial of the Cardio Flow FreedomFlow™ Orbital Atherectomy System to Treat Peripheral Artery Disease (FAST Trial) is a prospective non-randomized single arm study that will enroll up to 10 patients at 1 - 2 sites. The study will evaluate the safety and effectiveness of the Cardio Flow atherectomy device for plaque removal in de novo target lesions in the peripheral vasculature of the lower extremities. The primary safety endpoint is defined as freedom from a composite of new onset major adverse events through the 30-day follow-up as adjudicated by an independent Clinical Events physician. The primary effectiveness endpoint is defined as the ability of the Cardio Flow Device to achieve a residual diameter stenosis ≤ 50% without adjunctive therapy, determined by Angiographic core lab evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for percutaneous endovascular intervention in the lower extremity;
* Disease is located in peripheral arteries between 2mm and 5mm diameter;
* Ankle brachial index ≤ 0.90;
* Rutherford classification 2,3,4 or 5;
* De novo target lesion has ≥ 50% stenosis;
* Target lesion length ≤ 200 cm;
* At least 1 patent tibial vessel runoff;
* Written, signed informed consent.

Exclusion Criteria:

* Female not using adequate contraception or is breastfeeding;
* Rutherford class 0 1, and 6;
* target lesion within a native graft,
* in-stent restenosis,
* ≤ 50% occlusion, or chronic total occlusion;
* history of vascular surgery or interventional procedure on index limb within 30 days prior to procedure, or planned procedure within 30 days after index procedure, lesion in contralateral limb requiring intervention during index procedure or within 30 days of index procedure;
* known or suspected systemic infection;
* unstable coronary disease; significant kidney disease requiring dialysis;
* evidence of aneurysmal target vessel within past 2 months;
* evidence of intracranial or GI bleeding, intracranial aneurysm, MI or stroke within 2 months of baseline evaluation;
* history of heparin-induced thrombocytopenia;
* contraindication to anti-platelet, anticoagulant, or thrombolytic therapy;
* uncorrected bleeding disorders;
* thrombolytic therapy within 2 weeks of index procedure;
* life expectancy less than 12 months;
* unwilling or unable to comply with follow-up requirements;
* intraoperative complications due to the use of a marketed device prior to use of the atherectomy system;
* currently participating in an investigational drug or other device study that has not completed primary endpoint;
* unable to tolerate standard interventional procedures if the study device is not effective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Zang, MD, Study Director — Libra Medical
Locations (2):
- United States (2):
  - Cardiovascular Research of North Florida, LLC, Gainesville, Florida
  - Eastlake Cardiovascular, PC, Saint Clair Shores, Michigan

IPD SHARING:
Plan to Share IPD: No
Descriptive statistics of primary and secondary endpoints may be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Rutherford Classification [Mean (Standard Deviation); unit: units on a scale] — Rutherford Category is a number scale ranging from 0 to 6 with the following designation:
  0. Asymptomatic
  1. Mild claudication
  2. Moderate claudication
  3. Severe claudication
  4. Ischemic rest pain
  5. Minor tissue loss; nonhealing ulcer; local gangrene with diffuse pedal ischemia
  6. Major tissue loss extending above trans-metatarsal level
  units on a scale | 3.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treated Lesions With Achievement of ≤ 50% Residual Stenosis Without Adjunctive Therapy
Description: Achievement of ≤ 50% residual stenosis without adjunctive therapy as assessed angiographically on a per lesion basis
Time Frame: At time of procedure
Measure: Count of Units; unit: lesion
Units Other Than Participants: lesion
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Number analyzed (lesion) | 10
lesion | 3

2. Primary Outcome: Number of Participants Who Were Free From New-onset Major Adverse Events at 30 Days Post-treatment
Description: Major adverse events include the following:
  * All cause cardiovascular mortality.
  * Myocardial infarction (MI): Any newly diagnosed MI post procedure, defined as CK-MB ≥2X upper limit normal (ULN).
  * Clinically driven target lesion revascularization (TLR): any repeat percutaneous or surgical intervention to treat objectively documented symptoms of recurrent ischemia attributable to the treated lesion.
  * Clinically significant target vessel dissection: NHLBI grade C or greater as confirmed by angiography.
  * Clinically significant target vessel perforation: NHLBI Type III as confirmed by angiography.
  * Unplanned major target limb amputation: Amputation at the level of the trans-metatarsals or higher that was not previously planned
  * Clinically relevant distal embolization: Emboli requiring surgical or medical intervention and/or the presence of symptoms.
  * Pseudoaneurysm: disruption of the arterial wall at the treatment site as confirmed by angiography.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Participants | 10

3. Secondary Outcome: Serious Adverse Events
Description: All device and procedure related Serious Adverse Events at 30 days and 6 months
Time Frame: Through six months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Number of Lesions With Achievement of ≤ 50% Residual Stenosis With or Without Adjunctive Low-pressure Balloon Therapy
Description: Ability to achieve <50% residual diameter stenosis with or without adjunctive low-pressure balloon therapy on a per-lesion basis. Operator can follow atherectomy treatment with adjunctive balloon therapy.
Time Frame: At time of procedure
Measure: Count of Units; unit: Lesion
Units Other Than Participants: Lesion
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
Number analyzed (Lesion) | 11
Lesion | 11

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10)
Other (Gastrointestinal disorders) | 1 (1) — Patient scheduled for tracheostomy revision. Received a feeding tube and developed constipation.
Amputation below the knee (Infections and infestations) | 1 (2) — Left foot/toe pain due to gangrene with amputation of non-treated limb
Bleeding complication requires transfusion (Blood and lymphatic system disorders) | 1 (1) — GI bleed
Other (Infections and infestations) | 1 (4) — Non-healing wound treated with Vancomycin; Anemia requiring transfusion; acute kidney injury in setting of hyperglycemis treated with drugs
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10)
Other (Gastrointestinal disorders) | 1 (1) — Constipation
Other (Infections and infestations) | 1 (1) — Routine care visit revealed skin disorder. Treated with Bactrim DS
Other (Infections and infestations) | 1 (1) — Non-healing wound treated with Keflex
Other (Infections and infestations) | 1 (1) — Hepatitis C with hepatic steatosis. Discharged and referred to hepatoloogy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03365154/Prot_SAP_001.pdf
  • Informed Consent Form (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03365154/ICF_003.pdf